CLINICAL TRIAL: NCT06060548
Title: Role of a Novel Implantable Loop Recorder in the Management of Premature Ventricular Contractions
Brief Title: Role of Novel ILR in the Management of PVCs
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-ILR_PVC-0011
Record Dates: First submitted 2023-09-12; First posted 2023-09-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: PVC - Premature Ventricular Contraction; Myocarditis
MeSH Terms: conditions — Ventricular Premature Complexes; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with PVCs: Patients referred for management of symptomatic or asymptomatic PVCs. Patients presenting with PVCs and ventricular arrhythmias will be monitored using ILRs from the time of their initial presentation of PVCs.
  Interventions: Other: Monitoring of patients presenting with PVCs

INTERVENTIONS:
Other: Monitoring of patients presenting with PVCs — Patients presenting with PVCs and ventricular arrhythmias will be monitored using ILRs from the time of their initial presentation of PVCs to assess for the incidence of all cardiac arrhythmias. They will also be evaluated for clinical, biomarker and radiological evidence of myocarditis to understand association with incident arrhythmias.

SUMMARY:
This prospective, observational study is a single center clinical registry of patients referred for management of symptomatic or asymptomatic Premature Ventricular Contractions (PVCs). Subjects will be followed through 12 months. The study will enroll approximately 50 patients.

DETAILED DESCRIPTION:
This study is intended to monitor patients presenting with Premature Ventricular Contractions (PVCs) and ventricular arrhythmias using implantable loop recorders (ILRs) from the time of their initial presentation of PVCs to assess for the incidence of all cardiac arrhythmias detected with long term monitoring in this population. It is also intended to evaluate for clinical, biomarker and radiological evidence of myocarditis in this cohort to understand association with incident arrhythmias and understand the role of implantable loop recorders (ILRs)in managing these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Have a Medtronic LINQ II ILR
* Willing and able to give written informed consent

Exclusion Criteria:

* History of myocardial infarction
* Significant flow-limiting coronary artery disease (≥50% stenosis) on invasive coronary angiography or Computed tomography angiography (CTA).
* History of cardiac arrest
* With existing implantable defibrillators
* Currently pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred for management of symptomatic or asymptomatic PVCs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of unrecognized myocarditis | 12 Months
  Identification of unrecognized myocarditis in patients presenting PVCs with positive FDG-PET [fluorodeoxyglucose (FDG)-positron emission tomography (PET)] scanning.
Evaluation of efficacy of immunosuppressive therapy - PVC burden reduce | 12 Months
  Evaluation of efficacy of immunosuppressive therapy in patients with NICM with PVCs in reducing PVC burden as compared to their baseline PVC burden.
Evaluation of efficacy of immunosuppressive therapy - LVEF improvement | 12 Months
  Evaluation of efficacy of immunosuppressive therapy in patients with NICM by documenting improvement in LVEF compared to their baseline LVEF.
Associated atrial and ventricular arrhythmias | 12 Months
  Assessing incidence of associated atrial and ventricular arrhythmias as detected with ILR recordings in patients with apparently idiopathic PVCs.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (6):
- United States (6):
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn MS. Current Concepts of Premature Ventricular Contractions. J Lifestyle Med. 2013 Mar;3(1):26-33. Epub 2013 Mar 31. PMID 26064834
- [Background] Ng GA. Treating patients with ventricular ectopic beats. Heart. 2006 Nov;92(11):1707-12. doi: 10.1136/hrt.2005.067843. No abstract available. PMID 17041126
- [Background] Kennedy HL, Whitlock JA, Sprague MK, Kennedy LJ, Buckingham TA, Goldberg RJ. Long-term follow-up of asymptomatic healthy subjects with frequent and complex ventricular ectopy. N Engl J Med. 1985 Jan 24;312(4):193-7. doi: 10.1056/NEJM198501243120401. PMID 2578212
- [Background] Lakkireddy D, Turagam MK, Yarlagadda B, Dar T, Hamblin M, Krause M, Parikh V, Bommana S, Atkins D, Di Biase L, Mohanty S, Rosamond T, Carroll H, Nydegger C, Wetzel L, Gopinathannair R, Natale A. Myocarditis Causing Premature Ventricular Contractions: Insights From the MAVERIC Registry. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007520. doi: 10.1161/CIRCEP.119.007520. Epub 2019 Dec 16. PMID 31838913
- [Background] Ruberman W, Weinblatt E, Goldberg JD, Frank CW, Shapiro S. Ventricular premature beats and mortality after myocardial infarction. N Engl J Med. 1977 Oct 6;297(14):750-7. doi: 10.1056/NEJM197710062971404. PMID 70750
- [Background] Whiting RB. Ventricular premature contractions. Which should be treated? Arch Intern Med. 1980 Nov;140(11):1423-6. PMID 6159832
- [Background] Piccolo E, Raviele A. [Clinical and prognostic significance of hyperkinetic ventricular arrhythmias]. G Ital Cardiol. 1983;13(4):276-89. Italian. PMID 6350092
- [Background] Kastor JA. Ventricular premature beats. Adv Intern Med. 1983;28:63-91. PMID 6340432
- [Background] Wu AH. Management of patients with non-ischaemic cardiomyopathy. Heart. 2007 Mar;93(3):403-8. doi: 10.1136/hrt.2005.085761. No abstract available. PMID 17322525
- [Background] Tschope C, Cooper LT, Torre-Amione G, Van Linthout S. Management of Myocarditis-Related Cardiomyopathy in Adults. Circ Res. 2019 May 24;124(11):1568-1583. doi: 10.1161/CIRCRESAHA.118.313578. PMID 31120823
- [Background] Mattsson G, Magnusson P. Electrical storm in the inflamed heart: ventricular tachycardia due to myocarditis. Clin Case Rep. 2017 Jul 3;5(8):1327-1332. doi: 10.1002/ccr3.1071. eCollection 2017 Aug. PMID 28781852
- [Background] Te ALD, Wu TC, Lin YJ, Chen YY, Chung FP, Chang SL, Lo LW, Hu YF, Tuan TC, Chao TF, Liao JN, Chien KL, Lin CY, Chang YT, Chen SA. Increased risk of ventricular tachycardia and cardiovascular death in patients with myocarditis during the long-term follow-up: A national representative cohort from the National Health Insurance Research Database. Medicine (Baltimore). 2017 May;96(18):e6633. doi: 10.1097/MD.0000000000006633. PMID 28471960
- [Background] Kang M, Chippa V, An J. Viral Myocarditis. 2023 Nov 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459259/ PMID 29083732
- [Background] Frustaci A, Chimenti C. Immunosuppressive therapy in virus-negative inflammatory cardiomyopathy. Herz. 2012 Dec;37(8):854-8. doi: 10.1007/s00059-012-3694-x. PMID 23080270
- [Background] Chan AK, Dohrmann ML. Management of premature ventricular complexes. Mo Med. 2010 Jan-Feb;107(1):39-43. PMID 20222294
- [Background] Kindermann I, Barth C, Mahfoud F, Ukena C, Lenski M, Yilmaz A, Klingel K, Kandolf R, Sechtem U, Cooper LT, Bohm M. Update on myocarditis. J Am Coll Cardiol. 2012 Feb 28;59(9):779-92. doi: 10.1016/j.jacc.2011.09.074. PMID 22361396
- [Background] Fabre A, Sheppard MN. Sudden adult death syndrome and other non-ischaemic causes of sudden cardiac death. Heart. 2006 Mar;92(3):316-20. doi: 10.1136/hrt.2004.045518. Epub 2005 May 27. PMID 15923280